CLINICAL TRIAL: NCT01804023
Title: Comparison of Objective Biomarkers of Protocol Compliance and Product Adherence With Classic Markers of Compliance and Adherence
Brief Title: Biomarkers of Protocol Compliance and Product Adherence
Status: Completed | Type: Observational
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Other Study IDs: D13-125
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: HIV Prevention

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy women
  Interventions: Other: HEC placebo gel applicators

INTERVENTIONS:
Other: HEC placebo gel applicators — Participants will handle, but not insert, 4 applicators containing HEC placebo gel.
  Participants will vaginally insert and removed 8 applicators containing HEC placebo gel. Gel will be expelled in to the vagina from only 2 applicators.

SUMMARY:
The purpose of this study is to compare tests of vaginal insertion of applicators(visual inspection of returned applicators (VIRA), inspection of returned applicators under ultraviolet (UV) light, and DNA/protein markers) to determine which, if any, warrant use in a clinical trial of a new vaginal microbicide. The study will also determine whether indicators of semen can be detected on applicators and the degree to which they correlate with reported intercourse, and the correlation between vaginal bacteria detected by a vaginal swab and those detected from the applicator. In addition, the study will determine whether several factors that may be encountered in a clinical trial are likely to affect detection of these markers, including storage for 30 days vs. 7 days, wiping applicators after use, the presence of gel, and inter- and intra-woman variability. The study will also assess safety.

DETAILED DESCRIPTION:
Screening tests will be performed to detect exclusion criteria. After confirming the absence of point-of-care exclusion criteria, four applicators (#1 to 4, "sham" applicators) will be handled by the participant, but not inserted into the vagina and the gel will be expelled into a waste container. Four applicators (#5 to 8) will be inserted into the participant's vagina, one at a time, by the investigator, removed, and then the gel will be expelled into a waste container. Two applicators (#9 and 10) will be inserted into the participant's vagina, one at a time, and gel will be expelled into the participant's vagina. Finally, two applicators (#11 and 12) will be inserted into the participant's vagina, one at a time, by the investigator, removed and then the gel expelled into a waste container. Applicators #11 and 12 will then be wiped clean with a paper towel. Thus, each participant will provide a total of 12 applicators, half of which will be processed within one week of her visit and half of which will be processed in approximately one month of her visit. Three readers blinded to the status of the applicators (sham, inserted with or without gel expulsion) will determine, by VIRA and UV light assessment, whether or not the applicators were inserted vaginally. Additional laboratory personnel, who will also be blinded to the status of the applicators, will process the applicators for DNA and protein markers of product adherence and protocol compliance.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years old
* In good health, as evidenced by history
* No use of vaginal medications in the past 7 days
* At least 3 days from the end of their last menses
* Willing and able to comply with study procedures

Exclusion Criteria:

* Surgery or biopsy of the vagina or cervix within 30 days
* Have a history of a total hysterectomy (removal of the uterus and cervix)
* Pregnancy
* Positive buccal HIV test
* Other conditions that, in the opinion of the investigator, would constitute contraindications to participation in the study or would compromise the ability to comply with study protocols, such as any major chronic illness or a major psychiatric disorder (e.g., schizophrenia)
* Current participation in any other drug or device study, or any study which, in the opinion of the investigator, would jeopardize interpretation of results of this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, non-pregnant, HIV-uninfected women
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: VIRA | 7 days after insertion of vaginal applicators
Number of applicators on which Y chromosome-associated genes can be detected and degree of correlation between detection and the number of days since last penile/vaginal intercourse | 7 days after insertion of vaginal applicators
Degree of correlation of vaginal species obtained from vaginal applicators and vaginal species obtained from vaginal swabs | 7 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: VIRA | 30 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: UV Light Inspection | 7 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: UV Light Inspection | 30 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: DNA sequences of vaginal bacteria | 7 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: DNA sequences of vaginal bacteria | 30 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: Immunohistochemical tests for protein markers | 7 days after insertion of vaginal applicators
Sensitivity, specificity, PPV, and NPV of the following indicator of vaginal insertion: Immunohistochemical tests for protein markers | 30 days after insertion of vaginal applicators
Number of applicators on which Y chromosome-associated genes can be detected and degree of correlation between detection and the number of days since last penile/vaginal intercourse | 30 days after insertion of vaginal applicators
Degree of correlation of vaginal species obtained from vaginal applicators and vaginal species obtained from vaginal swabs | 30 days after insertion of vaginal applicators

SECONDARY OUTCOMES:
Difference in detection of these markers when applicators are processed within one week versus approximately 30 days after the participant's visit | 30 days after insertion of vaginal applicators
Difference in the sensitivity, specificity, NPV and PPV of detection of these markers when applicators are wiped off after removal from the vagina | 7 days after insertion of vaginal applicators
Difference in detection of these markers when gel is present, either from a current applicator insertion and gel expulsion or from previous and current applicator insertion and gel expulsion | 7 days after insertion of vaginal applicators
Difference in the sensitivity, specificity, NPV and PPV of detection of these markers when applicators are wiped off after removal from the vagina | 30 days after insertion of vaginal applicators
Difference in detection of these markers when gel is present, either from a current applicator insertion and gel expulsion or from previous and current applicator insertion and gel expulsion | 30 days after insertion of vaginal applicators

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Thurman, M.D., Principal Investigator — Clinical Research Center, Eastern Virginia Medical School, Norfolk, VA
Locations (1):
- Clinical Research Center, Eastern Virginia Medical School, Norfolk, Virginia, United States